CLINICAL TRIAL: NCT04890704
Title: Curcuminoids Can Prevent Contrast-induced Acute Kidney Injury in Chronic Kidney Disease Patients Undergoing Elective Coronary Procedures: A Randomized Controlled Trial
Brief Title: Curcuminoids and Contrast-induced Acute Kidney Injury
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 157/61
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Acute Kidney Injury; Contrast Media Toxicity; Curcuminoid; Chronic Kidney Diseases
Keywords: contrast-induced acute kidney injury; Curcuminoids; coronary angiography
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Diarylheptanoids

STUDY DESIGN:
Intervention Model Description: prospective, double-blinded, randomized placebo-controlled study
Who Masked: Investigator
Masking Description: stratified randomization and allocate concealment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumioids (Experimental): The investogators prescribed curcuminoids 1,500 mg/day . The regimen was curcuminoids 500 mg three times a day from three days before the procedure until two days after. All patients also received standard prophylaxis protocol which included 0.9% sodium chloride 1 mL/kg/hour, given 12 hours before and 12 hours after CAG unless contraindicated.
  Interventions: Drug: Curcuminoid
- Placebo (Placebo Comparator): The placebo was identical capsule given three times daily and the remaining protocols were the same as the active group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Curcuminoid — Patients were stratified according to baseline eGFR and diabetes status with 1:1 assignment into curcuminoids and placebo group. Curcuminoids (250 mg capsules) were purchased from the Government Pharmaceutical Organization of Thailand (Anti-ox® registration number 1A 1/60(H)), which contained curcumin: demethoxycurcumin: bis-demothoxycurcumin at the ratio of 1:0.5:0.2.
  Arms: Curcumioids
Drug: Placebo — Identical capsules were used for the placebo from the same manufacturer.
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate the role of curcuminoids in the prevention of CI-AKI in CKD patients.The result of the study was prophylactic administration with curcuminoids in addition to standard treatment reduce the incidence of CI-AKI CKD patients undergoing elective CAG.

DETAILED DESCRIPTION:
This study was a single-center, prospective, double-blinded, randomized placebo-controlled trial in CKD patients undergoing elective coronary angiography (CAG) at Vajira hospital from October 2018 to March 2019. Patients were stratified according to baseline estimate glomerular filtration rate (eGFR) and diabetes status. They were randomized to Curcuminoids 1,500 milligrams per day starting 3 days before and 2 days after coronary procedure or placebo. The primary outcome was the development of CI-AKI, defined as serum creatinine rising ≥ 0.3 mg/dL within 48 hours after coronary angiography. The secondary outcomes were overall AKI incidences within 7 days after CAG, changes in eGFR, IL-6 hs-CRP, and other adverse events.

A total of 60 patients were enrolled( 30 in curcuminoids group, and 30 in the control group). Overall AKI developed in 5 patients in control group and none in curcuminoids group (16.67% versus 0%, p-value 0.052). The results showed that curcuminoids could preserve changes in eGFR compared to the placebo group (-1.5 vs 2.5 mL/min/1.73m2, p-value <0.001 within 48 hours and -4 versus 1 mL/min/1.73m2, p-value 0.002 within 7 days). The high-sensitive C-reactive protein (hs-CRP) and IL-6 levels were not different between patients receiving curcuminoids and placebo. In curcuminoids group, 3 patients developed mild nausea and diarrhea that improved with supportive care. No serious adverse events were found in both groups.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing elective CAG at Vajira hospital from October 2018 to March 2019 were included in the study
* older than 18 years old
* stable eGFR 15-60 mL/min/1.73m2 in last 3 months.

Exclusion Criteria:

* dialysis-dependent
* post-kidney transplantation
* acute heart failure or critically ill
* history of contrast or turmeric allergy
* increasing of alanine aminotransferase (ALT) or alkaline phosphatase (ALP) more than three times of normal upper limits or post-cholecystectomy
* history of AKI (as evidence by sCr change ≥ 0.3 mg/dL) within 14 days before the study - using medication included NSAIDs, warfarin, immunosuppression, N-acetyl cysteine, ascorbic acid or contrast agents within 14 days before the study
* pregnancy or lactation o
* denied consent .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The incidence of AKI | 48 hours
  the incidence of CI-AKI development between the addition of curcuminoids to standard protocol and standard protocol alone in patients who underwent CAG

SECONDARY OUTCOMES:
AKI of any cause within seven days after CAG | 7 days
  The incidence overallof AKI form any causes
Change in eGFR | 0,7 days
  The final eGFR compared to baseline eGFR before CAG
Change in IL-6 and hs-CRP | 0.7 days
  The final levels of inflammatory markers at the completion of study compare to baseline
Adverse events | 7 days
  The adverse events of curcuminoids

CONTACTS AND LOCATIONS:
Locations (1):
- Navamindradhiraj University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
After pub

REFERENCES:
- [Result] Nash K, Hafeez A, Hou S. Hospital-acquired renal insufficiency. Am J Kidney Dis. 2002 May;39(5):930-6. doi: 10.1053/ajkd.2002.32766. PMID 11979336
- [Result] Mehran R, Dangas GD, Weisbord SD. Contrast-Associated Acute Kidney Injury. N Engl J Med. 2019 May 30;380(22):2146-2155. doi: 10.1056/NEJMra1805256. No abstract available. PMID 31141635
- [Result] Morcos R, Kucharik M, Bansal P, Al Taii H, Manam R, Casale J, Khalili H, Maini B. Contrast-Induced Acute Kidney Injury: Review and Practical Update. Clin Med Insights Cardiol. 2019 Nov 1;13:1179546819878680. doi: 10.1177/1179546819878680. eCollection 2019. PMID 31700251
- [Result] Kusirisin P, Chattipakorn SC, Chattipakorn N. Contrast-induced nephropathy and oxidative stress: mechanistic insights for better interventional approaches. J Transl Med. 2020 Oct 20;18(1):400. doi: 10.1186/s12967-020-02574-8. PMID 33081797
- [Result] Tasanarong A, Vohakiat A, Hutayanon P, Piyayotai D. New strategy of alpha- and gamma-tocopherol to prevent contrast-induced acute kidney injury in chronic kidney disease patients undergoing elective coronary procedures. Nephrol Dial Transplant. 2013 Feb;28(2):337-44. doi: 10.1093/ndt/gfs525. Epub 2013 Jan 12. PMID 23314316
- [Result] Weisbord SD, Gallagher M, Jneid H, Garcia S, Cass A, Thwin SS, Conner TA, Chertow GM, Bhatt DL, Shunk K, Parikh CR, McFalls EO, Brophy M, Ferguson R, Wu H, Androsenko M, Myles J, Kaufman J, Palevsky PM; PRESERVE Trial Group. Outcomes after Angiography with Sodium Bicarbonate and Acetylcysteine. N Engl J Med. 2018 Feb 15;378(7):603-614. doi: 10.1056/NEJMoa1710933. Epub 2017 Nov 12. PMID 29130810